CLINICAL TRIAL: NCT01931033
Title: An Open-Label Trial of Oxytocin in Adolescents With Autism Spectrum Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Gagan Joshi, Medical Director, Bressler Program for Autism Spectrum Disorders, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-P-001548
Record Dates: First submitted 2013-08-22; First posted 2013-08-29 (Estimated); Results first posted 2023-10-04 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Autism Spectrum Disorders; Pervasive Developmental Disorders; ASD; PDD
Keywords: Autism Spectrum Disorders; Pervasive Developmental Disorders; ASD; PDD; Oxytocin; Syntocinon; treatment
MeSH Terms: conditions — Autism Spectrum Disorder; Child Development Disorders, Pervasive | interventions — Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oxytocin (Experimental): Intranasal Oxytocin (brand name Syntocinon) will be administered daily (for a total daily dose of 48 IU) for 8 weeks.
  Interventions: Drug: Intranasal Oxytocin

INTERVENTIONS:
Drug: Intranasal Oxytocin
  Other Names: Syntocinon

SUMMARY:
This study is an 8-week open-label trial testing oxytocin nasal spray (Syntocinon) as a treatment for social impairment in adolescents with autism spectrum disorders (ASD). We hypothesize that oxytocin nasal spray will be safe, tolerable, and effective in improving the core symptoms of autism spectrum disorders in adolescents ages 11-17.

ELIGIBILITY:
Inclusion Criteria

1. Male and female outpatients ages 11-17 years
2. DSM-IV-TR PDD diagnosis of autistic disorder, Asperger's disorder, or PDD-NOS as established by clinical diagnostic interview and with the aid of the MGH ASD Symptom Checklist (MGH-ASD-SCL).
3. At least moderate severity of ASD impairment as measured by a raw score of ≥80 on the SRS and a severity score of ≥4 on CGI-PDD.
4. Participants and their parent/guardian must be able to speak and understand English sufficiently to comprehend the nature of the study and to allow for the completion of all study procedures required per protocol.
5. Subjects and their parent/guardian must be considered reliable reporters.
6. Each subject and their parent/guardian must understand the nature of the study and provide written informed assent/consent.
7. Subjects must be able to participate in mandatory blood draws.
8. Subjects with mood, anxiety, or disruptive behavior disorders will be allowed to participate in the study provided they do not meet any exclusionary criteria.

Exclusion Criteria

1. IQ <85
2. Total lack of spoken language
3. DSM-IV-TR PDD diagnosis of Rett's disorder or childhood disintegrative disorder.
4. Clinically unstable psychiatric conditions or judged to be at serious suicidal risk as determined by evaluating investigator.
5. History of substance use (except nicotine or caffeine) within past 3 months
6. Serious, stable or unstable systemic illness including hepatic, renal, gastroenterological, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic, immunologic, or hematologic disease.
7. Subjects with severe hepatic impairment (LFTs > 3 times ULN) and those with severely impaired renal function (eGFR < 30).
8. Pregnant or nursing females.
9. Known hypersensitivity to oxytocin.
10. Severe allergies or multiple adverse drug reactions.
11. A non-responder or history of intolerance to oxytocin, after treatment at adequate doses as determined by the clinician.
12. Subjects with significant nasal pathology (including atrophic rhinitis, recurrent nose bleeds, and history of hypophysectomy).
13. Investigator and his/her immediate family defined as the investigator's spouse, parent, child, grandparent, or grandchild.
14. Currently enrolled or recently participated (within the past 6 months) in a clinical trial of intranasal oxytocin.

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2013-10; Primary Completion 2016-02-22 (Actual); Study Completion 2016-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gagan Joshi, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants Ages 11-17: Participants ages 11-17 enrolled to receive oxytocin treatment
Period: Overall Study
Arm/Group | Participants Ages 11-17
Started | 8
Completed | 5
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Participants Ages 11-17
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 1
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in ASD Symptoms Social Responsiveness Scales 2 (SRS-2) Scales From Baseline to Week 8
Description: Change in ASD symptoms as measured by change from baseline on the Social Responsiveness Scale 2 (SRS-2) scale.
  The SRS-2 is a 65-item rating scale completed that is used to measure the severity of autism spectrum symptoms as they occur in natural settings. The SRS-2 School Age form is completed by a parent or guardian for patients ages 9-17 and the SRS-2 Adult Self-report is completed by patients ages 18-59. Total raw scores range from 0 to 195, with higher scores indicating increased symptom severity.
Time Frame: Week-8
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Participants Ages 11-17
Number analyzed (Participants) | 5
scores on a scale | -32.4 (17.25688)

2. Primary Outcome: Number of Participants With ≥30% Reduction in SRS Raw Score and CGI Improvement Scores of ≤ 2 at Week 8
Description: The SRS-2 is a 65-item rating scale completed that is used to measure the severity of autism spectrum symptoms as they occur in natural settings. The SRS-2 School Age form is completed by a parent or guardian for patients ages 9-17 and the SRS-2 Adult Self-report is completed by patients ages 18-59. Total raw scores range from 0 to 195, with higher scores indicating increased symptom severity. The Clinical Global Impression Improvement scale (CGI-ASD-I) is a clinician rated measure of ASD improvement. Improvement scores range from 1 (very much improved) to 7 (very much worse).
Time Frame: Week-8
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Ages 11-17
Number analyzed (Participants) | 5
Participants | 2

ADVERSE EVENTS:
Time Frame: 8 weeks (from baseline to end of study)
Arm/Group | Participants Ages 11-17
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 5/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants Ages 11-17 (N=8)
Nasal Irritation (General disorders) | 1 (2)
Restlessness (General disorders) | 1 (1)
Mental Fatigue (Psychiatric disorders) | 1 (5)
Anxiety (Psychiatric disorders) | 1 (1)
Headache (General disorders) | 1 (2)
Lump in Throat (General disorders) | 1 (1)
Tightness in Fingers (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No